CLINICAL TRIAL: NCT03677830
Title: Postoperative Pain Control & Relief in Neonates
Acronym: POPCORN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Involved investigators no longer at the investigating center
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Marya Strand, MD, Associate Professor of Pediatrics, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 29544
Record Dates: First submitted 2018-09-06; First posted 2018-09-19 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Pain, Postoperative; Premature Infant; Opioid Use
MeSH Terms: conditions — Pain, Postoperative; Premature Birth | interventions — Acetaminophen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The intervention (intravenous acetaminophen) and placebo (saline) will be distributed by the pharmacy and are visually indistinguishable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Acetaminophen (Active Comparator): Infants randomized to the intervention arm will receive scheduled IV acetaminophen per LexiComp dosing guideline (28 0/7-32 6/7 weeks 10 mg/kg/dose every 12 hours; 33 0/7-38 6/7 weeks 10 mg/kg/dose every 8 hours; >39 0/7 weeks 10 mg/kg/dose every 6 hours). N-PASS scores will guide administration of IV morphine. Continuous infusion of morphine will be started if an infant requires 3 doses of morphine within a 6-hour period and titrated as needed per N-PASS scores.
  Interventions: Drug: Acetaminophen
- Intravenous Placebo (Placebo Comparator): Infants randomized to the control arm will receive normal saline placebo IV at the appropriate volume and times for the gestational age. IV acetaminophen is concentrated at 10 mg/ml; corresponding saline volumes will be 1 ml to 5 ml, approximately, based on subject weight. Control infants will also have N-PASS scores assessed using the same protocol following the surgical procedure for 72 hours. Dosing of IV morphine will be the same as the dosing for the intervention arm.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Acetaminophen — Scheduled intravenous acetaminophen for post-operative pain to minimize opiate exposure.
  Other Names: Ofirmev 10 MG/ML Injectable Solution
  Arms: Intravenous Acetaminophen
Drug: Saline — Intravenous saline will be administered at appropriate volume and schedule for control group as a placebo.
  Arms: Intravenous Placebo

SUMMARY:
Pain control for newborns has made significant improvements over the last 30 years. The use of narcotics remains the standard of care for neonates undergoing minor and major surgeries. Narcotics, however, are associated with adverse effects such as respiratory depression, prolonged intubation and withdrawal symptoms. Acetaminophen (Tylenol©) has been proposed as an adjunct to reduce narcotic use but current evidence from well designed studies in newborns and premature infants is limited. This study will randomly assign neonates undergoing a surgery to either morphine plus acetaminophen or morphine alone for pain control. The subjects will be followed for 72 hours after the operation and evaluate the benefits of acetaminophen for pain control.

ELIGIBILITY:
Inclusion Criteria:

* All neonates ≥ 28 weeks of gestation and <44 weeks of gestation undergoing general surgery procedures (below) and managed postoperatively in the Neonatal Intensive Care Unit (NICU).

Minor procedures Inguinal hernia repair Laparoscopic or open gastrostomy tube placement Peritoneal drain placement for spontaneous intestinal perforation Gastroschisis bedside patch closure

Major procedures Laparoscopic or open Nissen fundoplication, duodenal atresia repair, Hirschsprung pull through, Ladd's procedure or excision of abdominal cyst Thoracoscopy or thoracotomy procedure Enterostomy or colostomy creation Exploratory laparotomy Revision or closure of enterostomy or colostomy Any Gastroschisis or omphalocele repair in operating room Repair or staged repair of congenital anorectal malformations Resection of sacrococcygeal teratoma

Exclusion Criteria:

* Any infant admitted with preoperative diagnosis of neonatal abstinence syndrome (NAS) or known intrauterine opiate exposure
* Any diagnosis of hepatitis exclusive of TPN-related biliary cholestasis
* Renal disease with creatinine >2.0 mg/dl at enrollment
* Intraventricular hemorrhage grade 3 or greater, or cerebellar hemorrhage
* Any patient with myotonic dystrophy or other congenital disease limiting validity of pain scoring
* Opiate exposure within 14 days of operative procedure
* Non-English-speaking parents/guardians

Max Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Total morphine exposure | 72 hours following surgical procedure
  Total amount of morphine received by infants for pain control post-operatively in mg/kg

SECONDARY OUTCOMES:
Total "as needed" morphine exposure | 72 hours following surgical procedure
  Total "as needed" or prn doses of morphine received by infants for pain control post-operatively in mg/kg

OTHER OUTCOMES:
Apnea of >20 seconds | 72 hours following surgical procedure
  Apnea episodes of >20 seconds documented by nursing staff after surgical procedure
Time to first feed | up to 2 weeks
  Number of hours to first enteral feeding after surgical procedure
Time to full enteral feeds | up to 8 weeks
  Number of hours/days until receiving all nutritional support enterally following surgical procedure
Time to endotracheal extubation | up to 2 weeks
  Number of hours from surgical procedure to endotracheal extubation
Incidence of opiate withdrawal symptoms | up to 8 weeks
  Number of infants that develop withdrawal symptoms from opiate exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Cardinal Glennon Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No